CLINICAL TRIAL: NCT03897231
Title: Prevalence of Non-adherence to Medication Among Patients on Chronic Hemodialysis - a Multicenter Cross-sectional Study
Brief Title: Prevalence of Non-adherence to Medication Among Patients on Chronic Hemodialysis
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Other Study IDs: NNF17OC0029778
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Medication Adherence; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Participants will be invited to participate in the study during their dialysis treatment at the participating hemodialysis outpatient centres. Allocated nurses at Copenhagen University Hospital, Rigshospitalet (MS, AB, LFH, AH), Copenhagen University Hospital, Hillerød (MPL) and Copenhagen University Hospital Herlev (TM) will be responsible for recruitment. Eligible patients will be informed orally and in writing about the study. Participants who wish to participate will be asked to provide informed consent and, following this, complete a paper-based questionnaire during treatment. Patients who have difficulty reading Danish and patients with visual or physical impairments that impinge on their ability to complete the questionnaires will be interviewed using a structured interview approach based on the questionnaires.

SUMMARY:
Background:

Non-adherence to medication among patients on chronic hemodialysis compromises treatment effects and results in increased morbidity, mortality and extensive costs to the healthcare system. To our knowledge, no studies have investigated the prevalence of non-adherence among Danish hemodialysis patients using a validated measure of non-adherence.

Aim:

The primary aim of this study was to investigate the prevalence of non-adherence among Danish patients on chronic hemodialysis measured by self-report.

Our second aim was to explore patients' beliefs about medicines and potential associations between beliefs and non-adherence to medication.

Our third aim was to explore the prevalence and severity of physical and emotional symptoms and potential associations with non-adherence to medication.

Design:

A multi-centre cross-sectional study according to the STROBE statement will be conducted from May 2019 - April 2021. The study will take place in the outpatient hemodialysis centres at three large University Hospitals in the Capital Region of Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of end stage kidney disease
* Must have received hemodialysis treatment ≥3 month at a hospital-based outpatient hemodialysis Centre
* Must be able to understand and speak Danish

Exclusion Criteria:

* cognitive impairment
* no current medication prescriptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage kidney disease receiving hemodialysis treatment ≥3 month at a hospital-based outpatient hemodialysis Centre in the Capital region of Denmark
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
the Morisky-Green-Levine scale (MAQ) | up to 8 months
  number of participants with non-adherence to medication assessed by scores of ≥1 indicating non-adherence
Medication adherence report scale (MARS) | up to 8 months
  number of participants with non-adherence to medication assessed by scores of less than 25 points indicating non-adherence

SECONDARY OUTCOMES:
Beliefs about medicines (BMQ) | up to 8 months
  number of participants that believe the necessity of their medication outweighs the cost of taking it assessed by scores ranging fra - 20 to + 20, with a postivie number indicating that patients belief in the benefit of mediciations overweights concerns about taking them
Dialysis symptom index | up to 8 months
  the overall symptom burden assessed by the total number of symptoms reported by each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-rasmussen, Professor, Principal Investigator — Department of Nephrology, Rigshospitalet
Locations (1):
- Department of Nephology, Copenhagen, Denmark

REFERENCES:
- [Derived] Mechta Nielsen T, Marott T, Hornum M, Feldt-Rasmussen B, Kallemose T, Thomsen T. Non-adherence, medication beliefs and symptom burden among patients receiving hemodialysis -a cross-sectional study. BMC Nephrol. 2023 Oct 27;24(1):321. doi: 10.1186/s12882-023-03371-3. PMID 37891566